CLINICAL TRIAL: NCT06035926
Title: Survey of Symptoms After a COVID Vaccination in Employees: a Retrospective Study.
Brief Title: Survey of Symptoms After a COVID Vaccination in Employees
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: EC number: 34-326 ex 21/22
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Symptoms Recoding SARS-CoV-2 After Vaccination
Keywords: SARS-CoV-2; Symptoms
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire

SUMMARY:
Background:

SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) has had us firmly in its grip for more than two years. In January 2021, the quality and risk management unit of the LKH (Landeskrankenhaus) -Univ. Klinikum Graz commissioned to carry out vaccinations for employees and subsequently for high-risk patients.

In the vaccination line, which was open for 85 days in 2021/22, the vaccines from Astra Zeneca, Biontech-Pfizer and Moderna were vaccinated. There were hardly any complications. The primary immunization, booster vaccination and booster vaccination were carried out.

Despite the small number of incidents in the sense of an immediate reaction, there were numerous sick leave.

Methods:

For this reason, in the course of the booster vaccination, starting from October 2021 to January 2022, every vaccinated person was asked to fill out a questionnaire. Participation was voluntary and was supported by the works councils of the Medical University and the LKH-University clinic Graz approved. The survey served to retrospectively record how many employees developed symptoms in response to the respective vaccination.

With this approach it will be possible to subject the responses to an in-depth statistical analysis in order to obtain a data-based contribution to the side effects of vaccines categorized with different vaccination schemes.

ELIGIBILITY:
Inclusion Criteria:

* Employees with appropriate indication (>4 months after the second vaccination) according to the recommendations of the national vaccination committee.
* Signed vaccination information sheet.

Exclusion Criteria:

* no booster vaccination.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Employees of the University Clinic Graz who get a booster vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 1093 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of symptoms after the respective vaccination | 10 Minutes
  Occurence of symptoms, assessed by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schwarz-Martelanz CM, Hoffmann M, Wedrich A, Berghold A, Reininghaus E, Reinisch S, Borenich A, Sendlhofer G. Vaccine side effects after vaccination against COVID-19 in employees at an University Hospital in Austria. Sci Rep. 2025 Nov 21;15(1):41353. doi: 10.1038/s41598-025-25329-1. PMID 41272132